CLINICAL TRIAL: NCT03443011
Title: Diagnostics in Diverticulitis (DIDit)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Centrallasarettet Västerås (Other); Mora Hospital, Landstinget Dalarna (Unknown)
Responsible Party: Principal Investigator, Arnar Thorisson, Consulting radiologist, Uppsala University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Dnr 2016/411
Record Dates: First submitted 2016-12-26; First posted 2018-02-22 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (Experimental): All participants will be examined with both CT techniques. First a low dose CT without intravenous contrast followed by the standard method, a full dose CT with intravenous contrast
  Interventions: Radiation: Low dose CT without intravenous contrast

INTERVENTIONS:
Radiation: Low dose CT without intravenous contrast — participants will receive an extra radiation dosage of about 3 milli Sievert (mSv) depending on patients height and weight. This is the radiation amount from the low dose CT protocol without intravenous contrast.

SUMMARY:
This study focuses on if low dose CT without intravenous contrast has a high enough specificity and sensitivity for acute diverticulitis that it can be used as the primary diagnostic method instead of a full dose CT with intravenous contrast which is the standard method in Sweden.

DETAILED DESCRIPTION:
Patients will be recruited from the emergency departments in Mora and Vastmanland hospitals. All patients over the age of 50 with clinically suspected acute diverticulitis that meet inclusions criterium will be asked for participation. A Clinical examination and blood samples will be drawn.

Subjects will be sent to the radiology department where they will undergo computed tomography (CT) of the abdomen. The CT protocol consists of a low dose non contrast enhanced CT followed by a normal dose CT with intravenous contrast. This is needed as randomization of patients is not possible due to the fact that the Clinical diagnosis of diverticulitis is difficult and unreliable. This would lead to the situation that we would not know if a participant in the low dose CT Group has diverticulitis which was not seen with the low dose protocol or if the patient did not have diverticulitis.

The radiologist on call will examine the full dose CT examination and write a report as routine. At a later date Three blinded radiologists will examine first all low dose CT examinations and grade them according to our CT protocol. At a later date the radiologists will evaluate all full dose CT examinations using the same CT protocol.

Findings will then be compared between the two different CT methods and sensitivity and specificity for low dose CT will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 50
* Clinically suspected acute diverticulitis
* Low abdominal pain
* WBC over 10 x 109/L or raised C-reactive protein levels 25 mg/L

Exclusion Criteria:

* Pregnancy
* Previous allergy to intravenous contrast
* Renal failure or other reasons that the patient cannot undergo CT with iv contrast
* Unable to give informed consent
* Dementia
* Language barrier

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Presence of diverticulitis on low dose CT and/or full dose CT | Baseline
  Colonic wall thickening >5mm, pericolic fat stranding and diverticula on CT

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Smedh, Professor, Study Director — Center for Clinical Reasearch Vasteras
Locations (1):
- Region Vastmanland Hospital, Västerås, Västmanland County, Sweden

IPD SHARING:
Plan to Share IPD: No